CLINICAL TRIAL: NCT02063516
Title: Comparison of Clinical Performance of the Guardian Laryngeal Mask With LMA Proseal - A Perspective, Randomized，Blind Study
Brief Title: Comparison of Clinical Performance of the Guardian Laryngeal Mask With LMA Proseal
Acronym: Guardian
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Haiyun Wang, vice-Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Wang001
Record Dates: First submitted 2014-01-13; First posted 2014-02-14 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2014-12

CONDITIONS: Efficacy of Oropharyngeal Seal Pressure
Keywords: Airway Cuff; Guardian; Proseal; Cuff Pressure; laryngeal Mask Airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guardian (Experimental): Device: Guardian Laryngeal Mask
  Interventions: Device: Guardian Laryngeal Mask
- Proseal (Experimental): Device:Proseal Laryngeal Mask Airway
  Interventions: Device: Proseal Laryngeal Mask Airway

INTERVENTIONS:
Device: Guardian Laryngeal Mask — Guardian Laryngeal Mask: The Guardian Laryngeal Mask (Ultimate Medical Pty Ltd, Richmond, Vic, Australia) is a new silicone-based single-use extraglottic airway device that forms a seal with the glottis for ventilation and with the hypopharynx for airway protection, and provides a gastric drainage port. In addition, it has a port for suctioning material from the hypopharynx and a pilot balloon valve that constantly monitors intracuff pressure. In the following randomized, non-crossover study, the investigators test if oropharyngeal leak pressures differed between the Guardian Laryngeal Mask and the LMA proseal in paralysed, anaesthetised patients.
  Arms: Guardian
Device: Proseal Laryngeal Mask Airway — Proseal Laryngeal Mask Airway: Silicon based, reusable, modified dorsal cuff and drainage tube
  Arms: Proseal

SUMMARY:
To compare insertion characteristics of 2 different supraglottic devices (Guardian LMA and Proseal LMA) and to observe any associated complications.

DETAILED DESCRIPTION:
Condition:

The study focuses on the comparison of the ease of insertion, oropharyngeal leak pressure, fiberoptic position and ease of gastric tube placement between the Guardian LMA and the LMA Proseal in paralyzed, anesthetized patients.

Device: Guardian Laryngeal Mask Device: LMA Proseal

Study Type:

Interventional

Study Design:

Allocation: Randomized Endpoint Classification: Efficacy Study Intervention Model: Parallel Assignment Masking: Single Blind (Subject)

ELIGIBILITY:
Inclusion Criteria:• Ambulatory patients scheduled to undergo knee arthroscopy, transurethral resection of bladder tumor, hand, gynecological and general surgical under a short general paralysed anesthesia of less than 2 hours (American Society of Anesthesiologists physical status I-II)

* 18 to 65 years of age
* Mallampati score less than 3
* thyromental distance more than 6.5 cm
* mouth opening more than >2.5 cm
* a body mass index less than 35 kg/m2;

Exclusion Criteria:

* Body weight 50 Kg
* Pregnancy
* Difficult airway
* Recent history of upper respiratory tract infection and sore throats
* A history of esophageal reflux disease
* ENT surgery
* Laparoscopic surgery
* Inability to understand the Study Information Sheet and provide a written consent to take part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Pajiyar AK, Wen Z, Wang H, Ma L, Miao L, Wang G. Comparisons of clinical performance of Guardian laryngeal mask with laryngeal mask airway ProSeal. BMC Anesthesiol. 2015 May 1;15:69. doi: 10.1186/s12871-015-0039-3. PMID 25929558

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Guardian | Proseal
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guardian | Proseal | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Age group include age >18-<65 years
  years | 45.75 (13.58) | 45.20 (14.78) | 45.47 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 8 | 36
  Male | 12 | 32 | 44
Weight [Mean (Standard Deviation); unit: kilogram] | 61.65 (8.95) | 59.75 (4.72) | 60.70 (7.12)
Height [Mean (Standard Deviation); unit: cm] | 162.20 (4.86) | 160.30 (4.11) | 161.22 (4.54)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.38 (2.71) | 23.27 (1.85) | 23.32 (2.29)
Type of surgery [Number; unit: participants]
  Gynecology | 18 | 20 | 38
  Orthopedic | 10 | 8 | 18
  Urology | 6 | 8 | 14
  General Surgery | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Oropharyngeal Seal Pressure
Description: This will be measured over the full range of cuff volumes (0-40 ml) and at an intracuff pressure of 60 cm H2O.
Time Frame: 5 min
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Guardian | Proseal
Number analyzed (Participants) | 40 | 40
cmH2O | 32.36 (4.93) | 29.41 (4.33)
Statistical Analysis 1: Comparison: Guardian vs Proseal; It was calculated that 80 adult patients randomized from different surgical department would have 80% power to detect a difference in 2 point in mean. Sampling size was determined using 2 sided t-test (alpha=0.05); Test type: Superiority or Other; p = 0.04, t-test, 2 sided

2. Secondary Outcome: Anatomic Position
Description: This will be determined fiberscopically via the airway tube over the full range of cuff volumes and at an intracuff pressure of 60 cm H2O.
Time Frame: 5 min
Population: Fiber-optic scoring system:
  "1, clear view of vocal cord" "2, Only arytenoids visible" "3, Only epiglottis visible" "4, No laryngeal structures visible"
Measure: Number; unit: participants
Arm/Group | Guardian | Proseal
Number analyzed (Participants) | 40 | 40
participants
  1 | 17 | 14
  2 | 20 | 21
  3 | 2 | 3
  4 | 1 | 2
Statistical Analysis 1: Comparison: Guardian vs Proseal; Test type: Superiority or Other; p = 0.836, Chi-squared

3. Other Pre Specified Outcome: Amount of Air Added to Keep Cuff Pressure 60cmH20.
Description: The accuracy of the intrinsic cuff pressure indicator is assessed by documenting which colour band the indicator is displaying when inflated according to manufacturers instructions, and measuring the numeric cuff pressure at the same time with a standard analogue cuff pressure gauge. The manufacturer has documented what pressure range is meant to be indicated by each of three colour ranges.
Time Frame: 30 minutes, 60 minutes, 90 minutes and 120 minutes
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Guardian | Proseal
Number analyzed (Participants) | 40 | 40
ml
  30 min | 1.34 (0.40) | 0.84 (0.15)
  60 min | 1.24 (0.30) | 0.86 (0.16)
  90 min | 1.34 (0.40) | 0.88 (0.17)
  120 min | 1.46 (0.44) | 0.96 (0.18)
Statistical Analysis 1: Comparison: Guardian vs Proseal; Amount of air added at 30 minutes to maintain cuff pressure 60cmH2O; Test type: Superiority or Other; p = 0.0035, t-test, 2 sided
Statistical Analysis 2: Comparison: Guardian vs Proseal; Amount of air added at 60 minutes to maintain cuff pressure 60cmH2O; Test type: Superiority or Other; p = 0.003, t-test, 2 sided
Statistical Analysis 3: Comparison: Guardian vs Proseal; Amount of air added at 90 minutes to maintain cuff pressure 60cmH2O; Test type: Superiority or Other; p = 0.0042, t-test, 2 sided
Statistical Analysis 4: Comparison: Guardian vs Proseal; Amount of air added at 120 minutes to maintain cuff pressure 60cmH2O; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1, 2 and 24 hours after the end of surgery
Description: The patients were asked 1, 2, and 24 hours after the end of surgery to assess post -operative complication. Sore throat was defined as " constant pain or discomfort in the throat independent of swallowing" ; dysphagia was defined as "difficulty or pain provoked by swallowing" ; dysphonia was defined as "difficulty or pain on speaking".
Arm/Group | Guardian | Proseal
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 10/40 | 12/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Guardian (N=40) | Proseal (N=40)
Sore throat (Injury, poisoning and procedural complications) | 6 | 7 — Sore throat was defined as " constant pain or discomfort in the throat independent of swallowing"
Dysphagia (Injury, poisoning and procedural complications) | 4 | 5 — difficulty or pain provoked by swallowing

LIMITATIONS AND CAVEATS:
We only use size-4 devices in adult patients with neuromuscular blockade, we presumed that same results would be obtained in patients who have not received neuromuscular blockade. lastly our data was not blinded causing potential source of bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No